CLINICAL TRIAL: NCT04286074
Title: Efficacy of a Physiotherapy Intervention by Training the Inspiratory Muscles With the Powerbreathe® Device to Improve Inspiratory Strength and Muscle Recovery in Semi-professional Soccer Players. A Randomized Clinical Study
Brief Title: Training of the Inspiratory Musculature in the Improvement of Inspiratory Strength and Muscle Recovery in Soccer Players
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Lockdown
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IMT
Record Dates: First submitted 2020-02-25; First posted 2020-02-26 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Breathing
Keywords: Breathing exercises; Soccer; Maximal respiratory pressures; Muscle Strength; Muscle fatigue
MeSH Terms: conditions — Respiratory Aspiration | interventions — multidrug resistance protein 50, Drosophila; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Each session will last 10 minutes, taking place 5 days a week, over a period of 6 weeks. The intervention will take place at the beginning of each training session.
  Prior to training, the muscle training technique will be performed against a resistance of 50% of the maximum inspiratory pressure of each athlete
  Interventions: Other: 50% resistance
- Control group (Active Comparator): Each session will last 10 minutes, taking place 5 days a week, over a period of 6 weeks. The intervention will take place at the beginning of each training session.
  Prior to training, the muscle training technique will be performed against a resistance of 10% of the maximum inspiratory pressure of each athlete
  Interventions: Other: 10% resistance

INTERVENTIONS:
Other: 50% resistance — Prior to training, the muscle training technique will be performed. The objective of applying the intervention using the Powerbreathe® device is to produce an increase in inspiratory force. The technique will be performed with the athlete standing, holding the device with his hand and his lips sealed on the mouthpiece. After a full expiration, you will make a quick and deep inspiration. The principal investigator of the study will ensure that the technique is performed correctly. There will be 2 series of 30 maximum inspirations. These interventions will be faced with a resistance of 50% of the maximum inspiratory pressure of each athlete
  Other Names: Experimental group
  Arms: Experimental group
Other: 10% resistance — Prior to training, the muscle training technique will be performed. The objective of applying the intervention using the Powerbreathe® device is to produce an increase in inspiratory force. The technique will be performed with the athlete standing, holding the device with his hand and his lips sealed on the mouthpiece. After a full expiration, you will make a quick and deep inspiration. The principal investigator of the study will ensure that the technique is performed correctly. There will be 2 series of 30 maximum inspirations. These interventions will be faced with a resistance of 10% of the maximum inspiratory pressure of each athlete
  Other Names: Control group
  Arms: Control group

SUMMARY:
Soccer requires the activation of aerobic and anaerobic metabolism. The increase of the ventilatory demand stimulates the increase of the neural impulse to the respiratory muscles, increasing the mechanical power of the inspiratory muscles.

The main objective of the study is to assess the effectiveness in the improvement of the strength of the inspiratory muscles and the muscular recovery with the Powerbreathe® device in semi-professional soccer players.

Randomized double-blind clinical study with follow-up period. 36 semi-professional soccer players from the province of Soria will be randomly distributed to the study groups: experimental (inspiratory muscle training with 50% resistance) and control (10% resistance training). The dependent variables will be: aerobic and anaerobic sports performance (Cooper's 12-Minute Run Test and Repeated Sprint Ability), blood lactate concentration (Lactate Scout®), and lung function using the ergo-respiratory parameters (maximum inspiratory pressure, expiratory pressure maximum, forced vital capacity and forced expiratory volume in 1 second). The sample distribution will be calculated using the Kolmogorov-Smirnov test. The changes after each evaluation will be analyzed with the t-student test and with an ANOVA of repeated measures, the intra and intersubject effect will be observed. The effect size will be calculated using Cohen's formula.

It is intended to observe improvement in inspiratory strength levels, decrease in blood lactate concentration and an increase in aerobic and anaerobic sports performance.

ELIGIBILITY:
Inclusion Criteria:

* Football players
* Male
* With an age range of 18 to 35 years
* Which currently compete in the category of Spanish third division nationally.

Exclusion Criteria:

* Subjects who have some type of injury that prevents them from practicing sports at the time of study
* With medical diagnosis of respiratory pathology
* That are not able to overcome the respiratory resistance of the device
* Have not signed the informed consent document.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline inspiratory force after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  An assessment will be made by spirometry of the maximum inspiratory pressure. A portable spirometer will be used (Mir Smart One model, MIR INC, New Berlin, WI, USA). The evaluation will be carried out according to the protocol indicated by the American Thoracic Society. The athlete will be placed in standing position holding the mouthpiece with his hand and with the wise sealed around it. After a full expiration you will proceed to a quick and deep inspiration. The unit of measure of this measuring instrument is cmH2O. A higher score indicates a greater inspiratory force.

SECONDARY OUTCOMES:
Change from baseline muscle recovery after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  It will be done by measuring blood lactate concentration. The measurement protocol used was described by Coyle et al. A puncture will be made in the earlobe for blood measurement, using puncture lancets, while the results will be analyzed with a lactate analyzer, model Lactate Scout 4 (model Scout Lactate, EKF Diagnostics, Germany). The unit of measure is mmol / l. A lower concentration of lactate in the blood indicates a greater capacity for muscle recovery.
Change from baseline aerobic performance after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  It will be done by applying the Cooper's 12-Minute Run test. With this test, the number of laps that the athlete is able to run in a period of 12 minutes, to an area of 300 meters, will be measured. The unit of measure is the number of turns that the player is able to perform, indicating a greater distance, a greater aerobic performance.
Change from baseline anaerobic performance after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  It will be done by applying the Repeated Sprint Ability (RSA) test. With this test, the time it takes for the athlete to make 6 sprints of 40 meters (20 + 20) with 20 seconds of rest between each one will be measured. The unit of measure is temporary (seconds). Performing sprints in less time indicates greater anaerobic performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain